CLINICAL TRIAL: NCT01037127
Title: An Open-Label, Multi-Center Study to Investigate the Objective Response Rate, Safety, and Pharmacokinetics of GSK1120212, a MEK Inhibitor, in BRAF Mutation-positive Melanoma Subjects Previously Treated With or Without a BRAF Inhibitor
Brief Title: Study to Determine the Effectiveness of GSK1120212 in BRAF Mutation-positive Melanoma Previously Treated With or Without a BRAF Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113583
Record Dates: First submitted 2009-11-25; First posted 2009-12-21 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-01

CONDITIONS: Cancer
Keywords: GSK1120212; BRAF Inhibitor; melanoma; MEK Inhibitor
MeSH Terms: conditions — Neoplasms; Melanoma | interventions — trametinib

ARMS (2):
- Cohort A (Experimental): Subjects who have had previous treatment with a BRAF inhibitor.
  Interventions: Drug: GSK1120212
- Cohort B (Experimental): Subjects who have had previous chemotherapy or immunotherapy without a BRAF inhibitor.
  Interventions: Drug: GSK1120212

INTERVENTIONS:
Drug: GSK1120212 — Daily oral dosing

SUMMARY:
MEK113583 is a Phase II open-label, multi-site study to investigate the objective response rate, safety, and pharmacokinetics of GSK1120212 in subjects with BRAF mutation-positive melanoma who were previously treated with or without a BRAF inhibitor. GSK1120212 is a potent and highly selective inhibitor of MEK activation and kinase activity.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic cutaneous melanoma that was previously treated with: (Cohort A) a BRAF inhibitor either with or without other prior therapy. (Cohort B) at least 1 prior chemotherapy or immunotherapy, without treatment with a BRAF inhibitor.
* Documented positive BRAF mutation (V600E, V600K, or V600D).
* Subjects must provide archived tumor tissue or undergo fresh tumor biopsy prior to enrollment.
* The subject must have a radiographically measurable tumor.
* The subject is able to carry out daily life activities without significant difficulty (ECOG performance status score of 0 or 1).
* Able to swallow and retain oral medication.
* Sexually active subjects must use acceptable methods of contraception during the course of the study.
* Adequate organ system function and blood cell counts.

Exclusion Criteria:

* The subject has had major surgery or received certain types of cancer therapy within 21 days before starting the study.
* Previous treatment with a MEK inhibitor.
* Current use of a prohibited medication listed in the protocol.
* Uncontrolled glaucoma.
* Brain metastasis, unless previously treated with surgery or stereotactic radiosurgery, and the disease has been stable for at least 2 months prior to enrollment.
* Current severe or uncontrolled systemic disease.
* History of clinically significant heart, lung, or eye/vision problems.
* Significant unresolved side effects from previous anti-cancer therapy.
* The subject is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- United States (6):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas
- Australia (3):
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, East Melbourne, Victoria
  - GSK Investigational Site, Nedlands, Western Australia

REFERENCES:
- [Result] Kim KB, Kefford R, Pavlick AC, Infante JR, Ribas A, Sosman JA, Fecher LA, Millward M, McArthur GA, Hwu P, Gonzalez R, Ott PA, Long GV, Gardner OS, Ouellet D, Xu Y, DeMarini DJ, Le NT, Patel K, Lewis KD. Phase II study of the MEK1/MEK2 inhibitor Trametinib in patients with metastatic BRAF-mutant cutaneous melanoma previously treated with or without a BRAF inhibitor. J Clin Oncol. 2013 Feb 1;31(4):482-9. doi: 10.1200/JCO.2012.43.5966. Epub 2012 Dec 17. PMID 23248257

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study used a 2-stage, Green-Dahlberg design that permitted stopping the trial for futility if <3 objective responses were observed in the first 30 participants enrolled. If >=3 objective responses were observed, 55 participants could be enrolled in each cohort.
Groups:
- Trametinib 2 mg: Prior BRAF Inhibitors: Participants who were previously treated (before the start of this study) with BRAF inhibitors received trametinib (GSK1120212) 2 milligram (mg) tablets orally once daily (qd) until treatment discontinuation criteria were met. Per the pre-specified study design, enrollment could have been stopped if objective response was observed in fewer than 3 participants among the first 30 participants enrolled. Per this criterion, enrollment in this cohort was stopped because, after enrollment of the first 30 participants, no objective responses were observed. Eligible participants who had been consented at the time the 30th participant was dosed were allowed to enroll, leading to overenrollment of 10 participants (total of 40 participants in this cohort). An interim analysis was performed after 30 participants had completed the first target post-dose disease assessment at 8 weeks.
- Trametinib 2 mg: Prior Standard Therapy: Participants who were previously treated with standard therapy, but not with BRAF inhibitors, received trametinib 2 mg tablets orally qd until treatment discontinuation criteria were met. Per the pre-specified study design, enrollment could have been stopped if objective response was observed in fewer than 3 participants among the first 30 participants enrolled. Per this criterion, 55 participants were enrolled in this cohort because objective responses occurred in 6 participants at the time of the interim analysis. Eligible participants who had been consented at the time the 55th participant was dosed were allowed to enroll. This led to the overenrollment of 2 participants (total of 57 participants in this cohort). An interim analysis was performed after 30 participants had completed the first target post-dose disease assessment at 8 weeks.
Period: Overall Study
Arm/Group | Trametinib 2 mg: Prior BRAF Inhibitors | Trametinib 2 mg: Prior Standard Therapy
Started | 40 | 57
Completed | 35 | 36
Not Completed | 5 | 21
Not completed — Lost to Follow-up | 2 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Study Closed Terminated | 2 | 17

BASELINE CHARACTERISTICS:
Groups:
- Trametinib 2 mg: Prior BRAF Inhibitors: Participants who were previously treated (before the start of this study) with BRAF (v-Raf murine sarcoma viral oncogene homolog B1) inhibitors received trametinib 2 milligram (mg) tablets orally once daily (qd) until treatment discontinuation criteria were met. Per the pre-specified study design, enrollment could have been stopped if objective response was observed in fewer than 3 participants among the first 30 participants enrolled. Per this criterion, enrollment in this cohort was stopped because, after enrollment of the first 30 participants, no objective responses were observed. Eligible participants who had been consented at the time the 30th participant was dosed were allowed to enroll, leading to overenrollment of 10 participants (total of 40 participants in this cohort). An interim analysis was performed after 30 participants had completed the first target post-dose disease assessment at 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Trametinib 2 mg: Prior BRAF Inhibitors | Trametinib 2 mg: Prior Standard Therapy | Total
Number analyzed (Participants) | 40 | 57 | 97
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.6 (14.52) | 54.0 (12.60) | 54.7 (13.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 25 | 43 | 68
Race/Ethnicity, Customized [Number; unit: Participants]
  White-Arabic/North African Heritage | 0 | 1 | 1
  White-White/Caucasian/European Heritage | 40 | 56 | 96

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Best Confirmed Response
Description: Best confirmed response was assessed by the Investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Best response was measured either as a complete response (CR), defined as the disappearance of all target lesions and pathological lymph nodes <10 millimeters (mm), or a partial response (PR), defined as at least a 30% decrease in the sum of the diameters of target lesions. To be assigned a status of confirmed CR or PR, a confirmatory disease assessment was required no less than 28 days after the criteria for response were first met.
Time Frame: From Baseline (Day 1) until the time of the first documented evidence of a confirmed complete response or partial response (up to approximately 25 weeks)
Population: All Treated Population: all participants who received at least one dose of investigational product
Measure: Number; unit: Participants
Groups:
- Trametinib 2 mg: Prior BRAF Inhibitors: Participants who were previously treated (before the start of this study) with BRAF inhibitors received trametinib 2 milligram (mg) tablets orally once daily (qd) until treatment discontinuation criteria were met. Per the pre-specified study design, enrollment could have been stopped if objective response was observed in fewer than 3 participants among the first 30 participants enrolled. Per this criterion, enrollment in this cohort was stopped because, after enrollment of the first 30 participants, no objective responses were observed. Eligible participants who had been consented at the time the 30th participant was dosed were allowed to enroll, leading to overenrollment of 10 participants (total of 40 participants in this cohort). An interim analysis was performed after 30 participants had completed the first target post-dose disease assessment at 8 weeks.
Arm/Group | Trametinib 2 mg: Prior BRAF Inhibitors | Trametinib 2 mg: Prior Standard Therapy
Number analyzed (Participants) | 40 | 57
Participants
  CR | 0 | 1
  PR | 0 | 13
Statistical Analysis 1: Comparison: Trametinib 2 mg: Prior Standard Therapy; Test type: Superiority or Other; percentage of participants = 25, 95% CI 2-sided [14.1 to 37.8] — The estimated value reflects the percentage of particpants with CR and PR

2. Primary Outcome: Number of Participants With Best Confirmed Response in the Indicated Subgroups of Participants Previously Treated With Standard Therapy But Not BRAF Inhibitors
Description: The number of participants with best confirmed response was analyzed for the following subgroups of participants previously treated with standard therapy but not BRAF inhibitors: (1) participants with prior (before the start of this study) brain metastases (mets); (2) participants without prior brain mets; (3) participants with BRAF mutation V600E; (4) participants with BRAF mutation V600E and no prior brain mets; and (5) participants with BRAF mutation V600K. Objective response was assessed per RECIST version 1.1. Objective response was measured either as CR, defined as the disappearance of all target lesions and pathological lymph nodes <10 mm, or PR, defined as at least a 30% decrease in the sum of the diameters of target lesions. To be assigned a status of confirmed CR or PR, a confirmatory disease assessment was required no less than 28 days after the criteria for response were first met. Brain metastasis is a cancer that has spread to the brain from another location of the body.
Time Frame: From Baseline (Day 1) until the time of the first documented evidence of a confirmed CR or PR (up to approximately 25 weeks)
Population: All Treated Population. A single participant could have been included in more than one subgroup. Subgroup analysis was not conducted in participants previously treated with BRAF inhibitors because there were no CRs or PRs among these participants.
Measure: Number; unit: Participants
Groups:
- Participants With Prior Brain Mets: Participants in this arm were those with prior (before the start of this study) brain metastasis, who were previously treated with standard therapy but not BRAF inhibitors. Participants received trametinib 2 mg tablets orally qd until treatment discontinuation criteria were met.
- Participants Without Prior Brain Mets: Participants in this arm were those without prior brain metastasis, who were previoulsy treated with standard thearpy but not BRAF inhibitors. Participants received trametinib 2 mg tablets orally qd until treatment discontinuation criteria were met.
- Participants With BRAF Mutation V600E: Participants in this arm were those with a positive BRAF mutation at V600E, who were previously treated with standard therapy but not with BRAF inhibitors. Participants received trametinib 2 mg tablets orally qd until treatment discontinuation criteria were met.
- Participants With BRAF Mutation V600E and no Prior Brain Mets: Participants in this arm were those with a positive BRAF mutation at V600E but no prior brain metastasis, who were previously treated with standard therapy but not with BRAF inhibitors. Participants received trametinib 2 mg tablets orally qd until treatment discontinuation criteria were met.
- Participants With BRAF Mutation V600K: Participants in this arm were those with a positive BRAF mutation at V600K, who were previously treated with standard therapy but not with BRAF inhibitors. Participants received trametinib 2 mg tablets orally qd until treatment discontinuation criteria were met.
Arm/Group | Participants With Prior Brain Mets | Participants Without Prior Brain Mets | Participants With BRAF Mutation V600E | Participants With BRAF Mutation V600E and no Prior Brain Mets | Participants With BRAF Mutation V600K
Number analyzed (Participants) | 12 | 45 | 46 | 36 | 8
Participants
  CR | 0 | 1 | 1 | 1 | 0
  PR | 2 | 11 | 11 | 9 | 0
Statistical Analysis 1: Comparison: Participants With Prior Brain Mets; Test type: Superiority or Other; percentage of participants = 17, 95% CI 2-sided [2.1 to 48.4] — The estimated value reflects the percentage of particpants with CR and PR
Statistical Analysis 2: Comparison: Participants Without Prior Brain Mets; Test type: Superiority or Other; percentage of participants = 27, 95% CI 2-sided [14.6 to 41.9] — The estimated value reflects the percentage of particpants with CR and PR
Statistical Analysis 3: Comparison: Participants With BRAF Mutation V600E; Test type: Superiority or Other; percentage of participants = 26, 95% CI 2-sided [14.3 to 41.4] — The estimated value reflects the percentage of particpants with CR and PR
Statistical Analysis 4: Comparison: Participants With BRAF Mutation V600E and no Prior Brain Mets; Test type: Superiority or Other; percentage of participants = 28, 95% CI 2-sided [14.2 to 45.2] — The estimated value reflects the percentage of particpants with CR and PR

3. Primary Outcome: Number of Participants With Best Unconfirmed Response at the Time of the Interim Analysis (Week 8)
Description: An interim analysis was performed using data collected approximately 12 and 13 weeks after the 30th participant was enrolled in the prior BRAF inhibitor and prior standard therapy groups, respectively. The best unconfirmed response by the investigator per RECIST version 1.1 was assessed. The study design permitted stopping the study for futility if <3 best confirmed responses were observed in the first 30 participants of each treatment arm after completing the first post-dose assessment at Week 8. Best response was measured as either a CR, defined as the disappearance of all target lesions and pathological lymph nodes <10 millimeters, or a PR, defined as at least a 30% decrease in the sum of the diameters of target lesions.
Time Frame: Week 8
Population: All Treated Population
Measure: Number; unit: Participants
Arm/Group | Trametinib 2 mg: Prior BRAF Inhibitors | Trametinib 2 mg: Prior Standard Therapy
Number analyzed (Participants) | 30 | 30
Participants
  CR | 0 | 0
  PR | 0 | 6
Statistical Analysis 1: Comparison: Trametinib 2 mg: Prior Standard Therapy; Test type: Superiority or Other; percentage of participants = 20, 95% CI [7.7 to 38.6] — The estimated value reflects the percentage of particpants with CR and PR

4. Secondary Outcome: Mean Plasma Concentrations
Description: Human plasma samples were analyzed for trametinib using a validated analytical method.
Time Frame: Day 15, pre-dose, 0.5-2 hours (hrs) post-dose, 2-4 hrs post-dose, and 4-8 hrs post-dose; Week 4, pre-dose; Week 8, pre-dose; Week 12, pre-dose
Population: Pharmacokinetic (PK) Population: all participants in the All Treated Population for whom PK samples were obtained and analyzed. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms (ng)/milliliter (mL)
Arm/Group | Trametinib 2 mg: Prior BRAF Inhibitors | Trametinib 2 mg: Prior Standard Therapy
Number analyzed (Participants) | 27 | 49
Nanograms (ng)/milliliter (mL)
  Day 15, pre-dose, n= 27, 44 | 12.3 (3.69) | 11.6 (5.54)
  Day 15, 0.5 to 2 hrs post-dose, n=23, 49 | 18.6 (7.23) | 15.2 (8.93)
  Day 15, 2 to 4 hrs post-dose, n=23, 48 | 23.6 (8.29) | 20.8 (9.87)
  Day 15, 4 to 8 hrs post-dose, n=22, 49 | 21.3 (6.14) | 19.0 (8.39)
  Week 4, pre-dose, n=23, 42 | 11.7 (3.82) | 11.6 (4.19)
  Week 8, pre-dose, n=19, 31 | 11.6 (4.67) | 11.8 (6.24)
  Week 12, pre-dose, n=7, 30 | 13.2 (3.75) | 12.5 (6.29)

5. Secondary Outcome: Number of Participants With Any Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a subject or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. AE and serious AE (SAE) data were collected from the start of the investigational product and continued until the End of Treatment Visit. Refer to the general Adverse AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From the date of the first dose of study medication until 28 days after the last dose (up to 477 days)
Population: All Treated Population
Measure: Number; unit: Participants
Arm/Group | Trametinib 2 mg: Prior BRAF Inhibitors | Trametinib 2 mg: Prior Standard Therapy
Number analyzed (Participants) | 40 | 57
Participants | 39 | 57

6. Secondary Outcome: Duration of Tumor Response
Description: Duration of tumor response is defined as the time from the first documented evidence of a CR or PR to disease progression (at least a 20 percent increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; unequivocal progression of non-target lesions, or the appearance of a new lesion) or death due to any cause. No participants who were previously treated with BRAF inhibitors had a CR, defined as the disappearance of all target lesions and pathological lymph nodes <10 millimeters, or a PR, defined as at least a 30% decrease in the sum of the diameters of target lesions; thus, no duration of response data can be presented.
Time Frame: From the time of the first documented evidence of a confirmed CR or PR until disease progression or death due to any cause (up to approximately 40 weeks)
Population: All Treated Population. Only those participants who had a confirmed CR or PR were analyzed for duration of response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trametinib 2 mg: Prior BRAF Inhibitors | Trametinib 2 mg: Prior Standard Therapy
Number analyzed (Participants) | 0 | 14
Months |  | 5.7 [3.7 to 9.2]

7. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the interval between the treatment start date and the earliest date of disease progression (at least a 20 percent increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; unequivocal progression of non-target lesions, or the appearance of a new lesion) or death due to any cause, whichever occurred first. Participants who had not progressed or died were censored at the date of the last adequate tumor assessment at the time of the cut-off.
Time Frame: Baseline (Day 1) until the time of disease progression or death due to any cause (up to approximately 57 weeks)
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trametinib 2 mg: Prior BRAF Inhibitors | Trametinib 2 mg: Prior Standard Therapy
Number analyzed (Participants) | 40 | 57
Months | 1.8 [1.8 to 2.0] | 4.0 [3.6 to 5.6]

8. Secondary Outcome: PFS in the Indicated Subgroups of Participants Previously Treated With Standard Therapy But Not BRAF Inhibitors
Description: PFS was analyzed for the following subgroups of participants previously treated with standard therapy but not BRAF inhibitors: (1) participants with prior (before the start of this study) brain metastases (mets); (2) participants without prior brain mets; (3) participants with BRAF mutation V600E; (4) participants with BRAF mutation V600E and no prior brain mets; and (5) participants with BRAF mutation V600K. Per RECIST version 1.1, PFS is defined as the interval between the treatment start date and the earliest date of disease progression (at least a 20 percent increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; unequivocal progression of non-target lesions, or the appearance of a new lesion) or death due to any cause, whichever occurred earliest. Brain metastasis is a cancer that has spread to the brain from another location of the body.
Time Frame: Baseline (Day 1) until the time of disease progression or death due to any cause (up to approximately 57 weeks)
Population: All Treated Population. A single participant could have been included in more than one subgroup. Subgroup analysis was not conducted in participants previously treated with BRAF inhibitors because this subgroup was stopped for futility and nearly all the participants progressed before 4 months.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Participants With Prior Brain Mets: Participants in this arm were those with prior (before the start of this study) brain metastasis who were previously treated with standard therapy but not with BRAF inhibitors received trametinib 2 mg tablets orally qd until treatment discontinuation criteria were met.
- Participants Without Prior Brain Mets: Participants in this arm were those without prior brain metastasis who were previously treated with standard therapy but not with BRAF inhibitors. Participants received trametinib 2 mg tablets orally qd until treatment discontinuation criteria were met.
- Participants With BRAF Mutation V600E: Participants in this arm were those with positive BRAF mutation at V600E, who were previously treated with standard therapy but not with BRAF inhibitors. Participants received trametinib 2 mg tablets orally qd until treatment discontinuation criteria were met.
- Paticipants With BRAF Mutation V600E and no Prior Brain Mets: Participants in this arm were those with positive BRAF mutation at V600E but no prior brain metastasis, who were previously treated with standard therapy but not with BRAF inhibitors. Participants received trametinib 2 mg tablets orally qd until treatment discontinuation criteria were met.
- Participants With BRAF Mutation V600K: Participants in this arm were those with positive BRAF mutation at V600K, who were previously treated with standard therapy but not with BRAF inhibitors. Participants received trametinib 2 mg tablets orally qd until treatment discontinuation criteria were met.
Arm/Group | Participants With Prior Brain Mets | Participants Without Prior Brain Mets | Participants With BRAF Mutation V600E | Paticipants With BRAF Mutation V600E and no Prior Brain Mets | Participants With BRAF Mutation V600K
Number analyzed (Participants) | 12 | 45 | 46 | 36 | 8
Months | 3.0 [1.8 to 5.3] | 4.6 [3.6 to 7.2] | 4.6 [3.6 to 5.7] | 5.3 [3.6 to 7.4] | 3.7 [1.8 to 4.6]

9. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the treatment start date until death due to any cause. Participants who had not died were censored at the date of the last adequate tumor assessment at the time of the cut-off.
Time Frame: Baseline (Day 1) until death due to any cause (up to 134 weeks)
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trametinib 2 mg: Prior BRAF Inhibitors | Trametinib 2 mg: Prior Standard Therapy
Number analyzed (Participants) | 40 | 57
Months | 5.5 [3.5 to 9.0] | 14.3 [11.3 to 24.4]

10. Secondary Outcome: Number of Participants Who Survived Until 6 Months, 12 Months and 24 Months From Baseline
Description: Overall survival (defined as the time from the treatment start date until death due to any cause) data data are presented as the number of participants who were alive 6 months, 12 months and 24 months after Baseline. Participants who had not died were censored at the date of the last adequate tumor assessment at the time of the cut-off.
Time Frame: Month 6, Month 12 and Month 24
Population: All Treated Population
Measure: Number; unit: Participants
Arm/Group | Trametinib 2 mg: Prior BRAF Inhibitors | Trametinib 2 mg: Prior Standard Therapy
Number analyzed (Participants) | 40 | 57
Participants
  Died at or prior to 6 months | 20 | 12
  Died after 6 months | 15 | 24
  Censored, less than 6 months follow-up | 3 | 1
  Censored, more than 6 months follow-up | 2 | 20
  Died at or prior to 12 months | 30 | 23
  Died after 12 months | 5 | 13
  Censored, less than 12 months follow-up | 3 | 1
  Censored, more than 12 months follow-up | 2 | 20
  Died at or prior to 24 months | 35 | 34
  Died after 24 months | 0 | 2
  Censored, less than 24 months follow-up | 3 | 2
  Censored, more than 24 months follow-up | 2 | 19

11. Secondary Outcome: Number of Participants With Tumor Progression
Description: Tumor progression was assessed as disease progression (DP), defined as at least a 20 percent increase in the sum of diameters of target lesions (representative of all involved organs), taking as reference the smallest sum on study; unequivocal progression of non-target lesions; or the appearance of a new lesion. Because melanoma often progresses to the brain/central nervous system (CNS) and this study enrolled approximately 20% participants with prior brain metastases, tumor progression in the brain/CNS was summarized. Paticipants could have been included in more than one category.
Time Frame: Baseline (Day 1) until tumor progression (up to approximately 57 weeks)
Population: All Treated Population
Measure: Number; unit: Participants
Arm/Group | Trametinib 2 mg: Prior BRAF Inhibitors | Trametinib 2 mg: Prior Standard Therapy
Number analyzed (Participants) | 40 | 57
Participants
  Number of participants (par.) with DP | 35 | 43
  Number of par. with DP in target lesions | 21 | 22
  Number of par. with DP in non-target lesions | 8 | 11
  Number of par. with a new lesion | 22 | 23
  Number of par. with clinical progression | 3 | 0

ADVERSE EVENTS:
Time Frame: Serious AEs and non-serious AEs are presented from the date of the first dose of study medication until the last participant's last visit (up to 1130 days).
Arm/Group | Trametinib 2 mg: Prior BRAF Inhibitors | Trametinib 2 mg: Prior Standard Therapy
Serious Adverse Events (participants affected / at risk) | 4/40 | 14/57
Other Adverse Events (participants affected / at risk) | 37/40 | 57/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trametinib 2 mg: Prior BRAF Inhibitors (N=40) | Trametinib 2 mg: Prior Standard Therapy (N=57)
Cellulitis (Infections and infestations) | 0 | 5
Pneumonia (Infections and infestations) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Blood amylase increased (Investigations) | 0 | 1
Cerebral hemorrhage (Nervous system disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Lipase increased (Investigations) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Pneumatosis (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Sepsis syndrome (Infections and infestations) | 0 | 1
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trametinib 2 mg: Prior BRAF Inhibitors (N=40) | Trametinib 2 mg: Prior Standard Therapy (N=57)
Rash (Skin and subcutaneous tissue disorders) | 20 | 32
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 8 | 21
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 20
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 17
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 8
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 4
Erythema (Skin and subcutaneous tissue disorders) | 2 | 6
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 5
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 3
Swelling face (Skin and subcutaneous tissue disorders) | 2 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 19 | 33
Nausea (Gastrointestinal disorders) | 19 | 23
Vomiting (Gastrointestinal disorders) | 11 | 16
Constipation (Gastrointestinal disorders) | 13 | 11
Abdominal pain (Gastrointestinal disorders) | 7 | 13
Dry mouth (Gastrointestinal disorders) | 8 | 6
Dyspepsia (Gastrointestinal disorders) | 4 | 4
Stomatitis (Gastrointestinal disorders) | 4 | 4
Abdominal distension (Gastrointestinal disorders) | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4
Flatulence (Gastrointestinal disorders) | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 4
Ascites (Gastrointestinal disorders) | 3 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 4
Mouth ulceration (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 14 | 24
Edema peripheral (General disorders) | 13 | 24
Pyrexia (General disorders) | 7 | 14
Face edema (General disorders) | 2 | 8
Chills (General disorders) | 3 | 7
Mucosal inflammation (General disorders) | 1 | 7
Pain (General disorders) | 1 | 4
Asthenia (General disorders) | 3 | 1
Cellulitis (Infections and infestations) | 4 | 3
Folliculitis (Infections and infestations) | 1 | 6
Localized infection (Infections and infestations) | 3 | 4
Urinary tract infection (Infections and infestations) | 5 | 3
Oral herpes (Infections and infestations) | 1 | 3
Postoperative wound infection (Infections and infestations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 10
Hypokalemia (Metabolism and nutrition disorders) | 3 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 | 4
Hyponatremia (Metabolism and nutrition disorders) | 4 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 5
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 8
Alanine aminotransferase increased (Investigations) | 1 | 6
Weight decreased (Investigations) | 2 | 5
Blood alkaline phosphatase increased (Investigations) | 2 | 1
Ejection fraction decreased (Investigations) | 0 | 4
Hemoglobin decreased (Investigations) | 2 | 1
Dizziness (Nervous system disorders) | 5 | 8
Headache (Nervous system disorders) | 3 | 5
Dysgeusia (Nervous system disorders) | 1 | 5
Neuropathy peripheral (Nervous system disorders) | 2 | 2
Vision blurred (Eye disorders) | 6 | 4
Eye edema (Eye disorders) | 2 | 0
Hypertension (Vascular disorders) | 0 | 12
Flushing (Vascular disorders) | 2 | 3
Lymphedema (Vascular disorders) | 3 | 2
Anemia (Blood and lymphatic system disorders) | 5 | 10
Insomnia (Psychiatric disorders) | 2 | 8
Depression (Psychiatric disorders) | 1 | 4
Mood altered (Psychiatric disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 0 | 3
Left ventricular dysfunction (Cardiac disorders) | 0 | 7
Breast enlargement (Reproductive system and breast disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 0 | 3
Visual impairment (Eye disorders) | 0 | 3
Skin fissures (Skin and subcutaneous tissue disorders) | 3 | 3
Hypoaesthesia (Nervous system disorders) | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 3
Sinus congestion (Infections and infestations) | 0 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Laceration (Injury, poisoning and procedural complications) | 0 | 3
Anxiety (Psychiatric disorders) | 2 | 1
Amnesia (Nervous system disorders) | 0 | 3
Hypotension (Vascular disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.